CLINICAL TRIAL: NCT02723513
Title: Bronchopulmonary Dysplasia: From Neonatal Chronic Lung Disease to Early Onset Adult Chronic Obstructive Pulmonary Disease
Brief Title: Bronchopulmonary Dysplasia: From Neonatal Chronic Lung Disease to Early Onset Adult COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Dr. Grace Parraga, PhD, Scientist, Robarts Research Institute, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ROB0041
Record Dates: First submitted 2016-03-19; First posted 2016-03-30 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Bronchopulmonary Dysplasia; Preterm Birth
Keywords: Proton MRI; Noble Gas MRI; Pulmonary Function
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preterm Adults (Experimental): All enrolled preterm adults will undergo non-contrast enhanced MRI (using ultra-short echo time methods), hyperpolarized noble gas MRI (using hyperpolarized xenon-129), x-ray computed tomography (CT), pulmonary function tests, and questionnaires in a single visit.
  Interventions: Other: Hyperpolarized Xenon-129

INTERVENTIONS:
Other: Hyperpolarized Xenon-129 — Hyperpolarized Xenon-129. Noble gas magnetic resonance imaging (MRI) has recently emerged as another research approach for the non-invasive measurement of lung structure and function, including conduction of gas through airways and into airspaces.
  Noble gas MRI provides a complimentary and alternative method for evaluating lung disease and may be superior to CT because it allows simultaneous visualization of both airway and airspace structure and function.

SUMMARY:
The investigators will apply xenon-129 (129Xe) and non-contrast enhanced magnetic resonance imaging (MRI) acquisition and analysis methods in 50 subjects aged between 20 and 29 years born pre-term (with and without a diagnosis of bronchopulmonary dysplasia [BPD]) and at term to characterize and probe the relationship between lung structure and function using imaging.

DETAILED DESCRIPTION:
This is a pilot, cross-sectional exploratory study to evaluate the relationship between imaging and other biomarkers in fifty patients born pre-term (with or without bronchopulmonary dysplasia [BPD]) and age-matched healthy controls. The term-born adults will serve as the controls.

All subjects will visit the Clinical Imaging Research Laboratories at Robarts Research Institute or the University of Montreal University Health Centre Sainte-Justine in a single visit and undergo: vital signs, pulmonary function testing (more specifically: spirometry, body plethysmography, airwave oscillation, and lung clearance index), questionnaires, proton and 129Xe MRI. Preterm patients will also have a low-dose chest computed tomography (CT), and have blood and urine samples taken for biomarkers of inflammation and oxidative stress.

MRI of the lungs will be performed using non-contrast enhanced methods (ultra-short echo time [UTE] MRI) and using an inhaled contrast agent: Hyperpolarized Xenon-129. Participants will inhale the hyperpolarized gas and perform a breathhold for up to 16 seconds. Four different types of images will be acquired in the coronal plain during each visit: 1) 1H thoracic cavity, 2) 129Xe static ventilation, 3) 129Xe diffusion weighted imaging, and, 4) multi-volume UTE MRI. Respiration and oxygen saturation will be monitored throughout the imaging session.

ELIGIBILITY:
Inclusion Criteria:

* 20-29 years old
* Pre-term (<29 weeks gestational age) with or without a diagnosis of bronchopulmonary dysplasia (BPD) or term born controls
* Subject understands the study procedures and is willing to participate in the study as indicated by the signature on the informed consent
* Subject is judged to be in otherwise stable health on the basis of medical history
* Subject is able to perform reproducible pulmonary function testing (i.e., the 3 best acceptable spirograms have FEV1 values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater)

Exclusion Criteria:

* Patient is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material
* Patient is unable to perform spirometry or plethysmography maneuvers
* Subject has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants)(at the discretion of the MRI Technologist/3T Manager)
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia
* Patient is pregnant

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with MRI-derived tissue signal intensity less than normal for age-matched individuals without BPD | Baseline
  This will be measured using non-contrast enhanced MRI methods (ultra-short echo time MRI) and hyperpolarized noble gas MRI methods. Mean whole lung signal intensity measurements will be quantified after the UTE MRI acquisition. Ventilation defect percent and apparent diffusion coefficients will be determined after noble gas MR acquisition.

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 s (FEV1) measured using spirometry | Baseline
Number of patients with abnormal Pulmonary Function measurement of surface-to volume ratio for gas exchange | Baseline
  diffusing capacity of carbon monoxide (DLCO) as a percent of predicted value for normal subjects of the same age and size

CONTACTS AND LOCATIONS:
Overall Officials: Grace Parraga, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada